CLINICAL TRIAL: NCT05102799
Title: MRI-phenotyping of Patients With Pathogenic Anoctamin 5 Variants
Acronym: ANO5 MRI
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Nanna Scharff Poulsen, Principal investigator, Rigshospitalet, Denmark
Other Study IDs: 1928485
Record Dates: First submitted 2021-10-20; First posted 2021-11-02 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Limb Girdle Muscular Dystrophy
Keywords: Anoctaminophathies
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Anoctaminopathies: Anoctaminopathies including Limb Girdle Muscular Dystrophy R12, Miyoshi distal Muscular Dystrophy type 3 and asymptomatic hyperCKemia
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
A large cohort of MRI scans from patients with pathogenic variants in the anoctamin 5 gene will be collected through an international collaboration to better describe muscle involvement.

DETAILED DESCRIPTION:
Background:

The anoctamin 5 gene (ANO5) encodes the anoctamine 5 protein that act as a calcium-sensitive chloride channel. The protein is preferentially expressed in skeletal and cardiac muscle and bone and likely acts in the repair of the cell membrane. Pathogenic ANO5 variants inherited in a autosomal recessive trait give rise to three main phenotypes: Limb-girdle muscular dystrophy type R12 (LGMDR12, formerly classified as LGMD2L), Miyoshi distal muscular dystrophy type 3 (MMD3), and asymptomatic hyperCKemia). As the name implies, patients with LGMDR12 are affected more proximally and patients with MMD3 more distally, but the definition and distinction between the two entities is unclear. Men with anoctaminopathy are more severely affected than women. Cardiac disease such as arrhythmias and cardiomyopathy as well as bulbar symptoms or respiratory failure are very rare in anoctaminopathies. Onset is in adulthood and disease progression is slow, generally with a later onset and disease progression than seen in other LGMDs. Ambulation is preserved until late in the disease course.

However, only few studies based on small case series have investigated the phenotype of patients with ANO5 mutations using MRI. There is therefore a need to investigate a larger international group of patients using MRI to properly describe which muscles are affected in men and women with anoctaminopathy.

The spectrum of phenotypes in anoctaminopathies resembles that seen in dysferlinopathies, and in the latter group, it has been shown that the former division into LGMDR2 (formally LGMD2B) and Miyoshi distal muscular dystrophy type 2 (MMD2) is rather arbitrary. Our hypothesis is that this may very well also be the case for LGMDR12 and MMD3. A large MRI study would be able to shed light on this question. Muscle involvement in patients with ANO5 mutations is said to be asymmetric based on clinical assessments (7,8,10). The proposed study will also elucidate this by studying symmetry of muscle affection. Finally, the diseases severity is said to be marked between the two sexes, but this has not been quantified in any detail before. The proposed study will also be able to shed light on this.

Aim:

The aims of the project are:

* To describe the muscle MRI phenotype in around 200 patients from multiple countries around the world.
* To investigate if it makes sense to group patients with pathogenic ANO5 variants into proximal and distal myopathies.
* To investigate to what extent the disease is asymmetric.
* To investigate the difference in disease severity between sexes.
* To investigate whether a phenotype-genotype correlation exists.

Methods:

Sites from all over the world will share an eCRF and their MRI data with Copenhagen Neuromuscular Center through the platform MyoShare.

ELIGIBILITY:
Inclusion Criteria:

* Two pathogenic variants in the anoctamin-5 gene
* T1-weighted MR-images of lower back and leg muscles.

Exclusion Criteria:

- Concomitant other disorders that also can result in muscular atrophy, i.e. polyneuropathy, other muscle diseases, recent long-term stay in intensive care, among others.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: MRIs of patients with pathogenic variants in the anoctamin 5 gene will be examined. The MRIs are obtained from either former studies or as part of clinical evaluation in the collaborating countries.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative fat fraction lower back and legs | 15 minutes
  Qualitative muscle fat fraction analyses of lower back and legs evaluated from T1-weighted images using the Mercury score (score: 0-4)

SECONDARY OUTCOMES:
Qualitative fat fraction of whole body | 15 minutes
  Qualitative fat fraction analyses of the rest of the body evaluated from T1-weighted images using the Mercury score (score: 0-4)
Quantitative fat fraction of axial and leg muscles | 60 minutes
  Qualitative fat fraction analyses of axial and leg muscles evaluated from Dixon images
Inflammatory evaluation of axial and leg muscles | 60 minutes
  Quantitative analysis of inflammation in axial and leg muscles from STIR images

CONTACTS AND LOCATIONS:
Locations (1):
- Nanna Scharff Poulsen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Little AA, McKeever PE, Gruis KL. Novel mutations in the Anoctamin 5 gene (ANO5) associated with limb-girdle muscular dystrophy 2L. Muscle Nerve. 2013 Feb;47(2):287-91. doi: 10.1002/mus.23542. Epub 2012 Nov 21. PMID 23169617
- [Background] Witting N, Duno M, Petri H, Krag T, Bundgaard H, Kober L, Vissing J. Anoctamin 5 muscular dystrophy in Denmark: prevalence, genotypes, phenotypes, cardiac findings, and muscle protein expression. J Neurol. 2013 Aug;260(8):2084-93. doi: 10.1007/s00415-013-6934-y. Epub 2013 May 14. PMID 23670307
- [Background] Palmio J, Penttila S, Jokela M. ANO5-Related Muscle Disease. 2012 Nov 29 [updated 2025 May 15]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK114459/ PMID 23193613
- [Background] Sarkozy A, Deschauer M, Carlier RY, Schrank B, Seeger J, Walter MC, Schoser B, Reilich P, Leturq F, Radunovic A, Behin A, Laforet P, Eymard B, Schreiber H, Hicks D, Vaidya SS, Glaser D, Carlier PG, Bushby K, Lochmuller H, Straub V. Muscle MRI findings in limb girdle muscular dystrophy type 2L. Neuromuscul Disord. 2012 Oct 1;22 Suppl 2:S122-9. doi: 10.1016/j.nmd.2012.05.012. PMID 22980763
- [Background] Ten Dam L, van der Kooi AJ, Rovekamp F, Linssen WH, de Visser M. Comparing clinical data and muscle imaging of DYSF and ANO5 related muscular dystrophies. Neuromuscul Disord. 2014 Dec;24(12):1097-102. doi: 10.1016/j.nmd.2014.07.004. Epub 2014 Aug 1. PMID 25176504
- [Background] Silva AMS, Coimbra-Neto AR, Souza PVS, Winckler PB, Goncalves MVM, Cavalcanti EBU, Carvalho AADS, Sobreira CFDR, Camelo CG, Mendonca RDH, Estephan EDP, Reed UC, Machado-Costa MC, Dourado-Junior MET, Pereira VC, Cruzeiro MM, Helito PVP, Aivazoglou LU, Camargo LVD, Gomes HH, Camargo AJSD, Pinto WBVDR, Badia BML, Libardi LH, Yanagiura MT, Oliveira ASB, Nucci A, Saute JAM, Franca-Junior MC, Zanoteli E. Clinical and molecular findings in a cohort of ANO5-related myopathy. Ann Clin Transl Neurol. 2019 Jul;6(7):1225-1238. doi: 10.1002/acn3.50801. Epub 2019 Jun 11. PMID 31353849
- [Background] Mahjneh I, Bashir R, Kiuru-Enari S, Linssen W, Lamminen A, Visser Md. Selective pattern of muscle involvement seen in distal muscular dystrophy associated with anoctamin 5 mutations: a follow-up muscle MRI study. Neuromuscul Disord. 2012 Oct 1;22 Suppl 2:S130-6. doi: 10.1016/j.nmd.2012.02.007. PMID 22980764
- [Background] Khawajazada T, Kass K, Rudolf K, de Stricker Borch J, Sheikh AM, Witting N, Vissing J. Muscle involvement assessed by quantitative magnetic resonance imaging in patients with anoctamin 5 deficiency. Eur J Neurol. 2021 Sep;28(9):3121-3132. doi: 10.1111/ene.14979. Epub 2021 Jul 11. PMID 34145687
- [Background] Willis TA, Hollingsworth KG, Coombs A, Sveen ML, Andersen S, Stojkovic T, Eagle M, Mayhew A, de Sousa PL, Dewar L, Morrow JM, Sinclair CD, Thornton JS, Bushby K, Lochmuller H, Hanna MG, Hogrel JY, Carlier PG, Vissing J, Straub V. Quantitative muscle MRI as an assessment tool for monitoring disease progression in LGMD2I: a multicentre longitudinal study. PLoS One. 2013 Aug 14;8(8):e70993. doi: 10.1371/journal.pone.0070993. eCollection 2013. PMID 23967145